CLINICAL TRIAL: NCT02240641
Title: Study on Protective Effect of Caldine® on Renal Function in Patients With a Balanced Hypertension
Brief Title: Effect of Caldine® on Renal Function in Balanced Hypertension
Status: Terminated | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 231.334
Record Dates: First submitted 2014-08-28; First posted 2014-09-16 (Estimated); Last update posted 2014-09-16 (Estimated); Status verified 2014-09

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — lacidipine; Diuretics; Antihypertensive Agents; Adrenergic alpha-Antagonists; Angiotensin-Converting Enzyme Inhibitors; Adrenergic beta-Antagonists

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- hypertension treatment strategies
  Interventions: Drug: Lacidipine; Drug: Diuretics; Drug: antihypertensive drugs; Drug: alpha blockers; Drug: Angiotensin-Converting Enzyme Inhibitors; Drug: beta blockers

INTERVENTIONS:
Drug: Lacidipine
  Other Names: Caldine
Drug: Diuretics
Drug: antihypertensive drugs
Drug: alpha blockers
Drug: Angiotensin-Converting Enzyme Inhibitors
Drug: beta blockers

SUMMARY:
The study aimed at comparing the evolution of renal function in patients showing a hypertension treated by various therapeutic strategies.

Due to the contract research organisation (CRO) decision in September 2000, the database was locked and not accessible for Boehringer Ingelheim France. Consequently it was decided to stop the study and not proceed to the analysis. Thus, only safety data were processed in the safety database.

ELIGIBILITY:
Inclusion Criteria:

* patients with hypertension requiring treatment

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with hypertension requiring treatment
Sampling Method: Non-Probability Sample
Enrollment: 5417 (Actual)
Dates: Start 1998-05; Primary Completion 2000-09 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events | up to two years